CLINICAL TRIAL: NCT05093712
Title: Patient-Informed Educational Intervention to Improve Cervical Cancer Literacy
Brief Title: Patient-Informed Educational Intervention for the Improvement of Cervical Cancer Literacy
Status: Withdrawn | Type: Observational
Why Stopped: Due to the limited resources and staffing needed in order to run the trial.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1269; NCI-2021-10696 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1269 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Stage IB Cervical Cancer FIGO 2018; Stage IB1 Cervical Cancer FIGO 2018; Stage IB2 Cervical Cancer FIGO 2018; Stage IB3 Cervical Cancer FIGO 2018; Stage II Cervical Cancer FIGO 2018; Stage IIA Cervical Cancer FIGO 2018; Stage IIA1 Cervical Cancer FIGO 2018; Stage IIA2 Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018; Stage III Cervical Cancer FIGO 2018; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IIIC Cervical Cancer FIGO 2018; Stage IIIC1 Cervical Cancer FIGO 2018; Stage IIIC2 Cervical Cancer FIGO 2018; Stage IVA Cervical Cancer FIGO 2018
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I (survey): Patients complete surveys over 10 minutes on their background, health literacy level, barriers to cancer care, and knowledge of cervical cancer and its treatment.
  Interventions: Other: Survey Administration
- Phase II (survey, educational video): Patients watch educational video on cervical cancer. Patients also complete surveys over 5-10 minutes at baseline and after watching educational video.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Watch educational video
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Groups: Phase II (survey, educational video)
Other: Survey Administration — Complete surveys

SUMMARY:
This study investigates the health literacy, cervical cancer knowledge, and radiation knowledge of patients with cervical cancer. The goal of this study is to develop a video that can improve patients 'understanding of cervical cancer and its treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the baseline health literacy, cervical cancer knowledge and radiation knowledge in a diverse sample of patients from two hospitals in Houston, Texas. (Phase 1) II. To test improvement in comprehension of cervical cancer and radiation terminology in a diverse sample of cervical cancer patients after viewing the video-based educational tool developed in this study. (Phase 2)

SECONDARY OBJECTIVES:

I. To assess barriers to care and assess baseline radiation adherence, defined as missing no treatments and time to radiation completion, in a diverse sample of patients from two hospitals in Houston, Texas.

II. To describe the impact of the video on radiation treatment adherence in terms of radiation completion, defined as missing no treatments) and time to radiation completion.

III. To describe the relationships between time to radiation completion, health literacy, sociodemographics, reported barriers to care, and baseline cervical cancer knowledge and misconceptions.

OUTLINE:

PHASE I: Patients complete surveys over 10 minutes on their background, health literacy level, barriers to cancer care, and knowledge of cervical cancer and its treatment.

PHASE II: Patients watch educational video on cervical cancer. Patients also complete surveys over 5-10 minutes at baseline and after watching educational video.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven carcinoma of the cervix
* Federation of Gynecology and Obstetrics (FIGO) stage IB-IVA
* N0 and N1 nodal status according to TNM staging
* Planned for definitive chemoradiation with curative intent
* Able to speak and read English or Spanish
* Age 18 or older
* Able to give informed consent

Exclusion Criteria:

* Physicians or nurses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women from MD Anderson Cancer Center and Harris Health System's Smith Clinic with biopsy proven carcinoma of the cervix
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Health literacy (Phase I) | Baseline
  The proportion of patients answering a particular knowledge item correctly will be calculated along with 95% score confidence intervals. As part of a secondary set of analyses, the percent of knowledge items answered correctly will be tabulated for each participant. Descriptive statistics and 95% confidence intervals will be calculated for percent of items answered correctly, both by site and combining data from both sites.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Klopp, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org